CLINICAL TRIAL: NCT05407480
Title: Therapeutic Recommendations for Children Registered in the RFAOP Register and With a Hodgkin Lymphoma
Brief Title: Thereapeutic Recommendantion for Children With a Hodgkin Lymphoma
Acronym: GFAOPLH2019
Status: Recruiting | Type: Observational
Sponsor: French Africa Pediatric Oncology Group (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: GFAOP LH 2019
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Staging; Therapeutic Recommendations
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational — Descriptive data will be collected to evaluation compliance with the protocol and to evaluate outcome

SUMMARY:
The GFAOP propose a simple and reproducible staging according to clinical, biological and radiological data.

Develop standardized but different therapeutic recommendations based on the availability or lack of radiation therapy in the pilot unites who will adapt these recommendations.

DETAILED DESCRIPTION:
In high-income countries, therapeutic outcomes exceed 90% and therapeutic de-escalation is necessary to reduce mainly the effects of long-term radiotherapy. Within the same country, there are also differences between the therapeutic protocols used in the different centres.

The Experience of Sub-Saharan African Units of the Franco-African Paediatric Oncology Group (GFAOP) in the treatment of pediatric Hodgkin lymphoma in 104 patients was based on chemotherapy alone. The latter was based on COPP/ABV cures without complementary irradiation adapted to the initial stratification and modulated according to the morphological response. Overall survival at 5 years was 82% at 30 months after a median decrease of 17 months.

It seemed appropriate to bring together in a single committee the representatives of the various pilot units in order to standardize the therapeutic protocols in the African countries.

So with this recommendation the GFAOP propose a simple and reproducible staging according to clinical, biological and radiological data.

- Develop standardized but different therapeutic recommendations based on the availability or lack of radiation therapy in the pilot unit.

ELIGIBILITY:
Inclusion Criteria:

under 18 years of age at diagnosis

* suffering from "classical" Hodgkin's disease according to the WHO classification.
* with no history of hematological malignancies or constitutional or acquired immune deficiencies

Exclusion Criteria:

* Over 18 years of age at diagnosis
* A history of hematological malignancies or a history of constitutional or a history of acquired immune deficiencies

Ages: 0 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children arriving in one of the participating units :
  under 18 years of age at diagnosis and suffering from "classical" Hodgkin's disease according to the WHO classification.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2034-11-20 (Estimated)

PRIMARY OUTCOMES:
Patient status | 24 months
  Dead or Alive
Drugs | 24 months
  The evaluation of the number of children who remain untreated because of lack of acess to chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: FATEN Ben Ayed, Professeur, Principal Investigator — French Africa Pediatric Oncology Group
Locations (1):
- Brenda Mallon, Paris, France, France

IPD SHARING:
Plan to Share IPD: No